CLINICAL TRIAL: NCT00726219
Title: Influence of the Insertion Distance on Loss of Sensation Produced by Femoral Perineural Catheters in the Context of Major Knee Surgery.
Brief Title: Insertion Distance of Femoral Perineural Catheters in the Context of Major Knee Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Dr Stephan Williams, Centre Hospitalier de l'Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD07.052
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2010-06

CONDITIONS: Total Knee Arthroplasty
Keywords: Major; knee; surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Insertion distance of femoral catheter: 3cm
  Interventions: Other: Femoral perineural catheter
- 2 (Other): Insertion distance of femoral catheter: 7cm
  Interventions: Other: Femoral perineural catheter

INTERVENTIONS:
Other: Femoral perineural catheter — Comparison of 2 insertion distances (3 vs 7 cm) for a femoral perineural catheter in the context of major knee surgery.

SUMMARY:
This study is designed to compare femoral perineural catheter insertion distances, in order to help determine which is the best for pain relief after knee surgery.

Hypothesis: the quality of the femoral nerve block will not be inferior if the catheter is inserted deeper (7cm compared to 3 cm)

DETAILED DESCRIPTION:
Pain after knee surgery is reported as severe for 60% of patients, and is a major concern in both hospitalised and ambulatory surgery patients. Pain control is particularly important, as adequate analgesia allows rapid mobilisation of the operated knee and prevents complications related to immobility. Several methods have been proposed to treat this pain, the most promising being injection of local anesthetic close to the femoral nerve. The injection of local anesthetics around the femoral nerve reduces sensation from the knee and provides better pain relief after surgery than narcotic medication. To prolong the duration of the analgesia, a small catheter must be positioned next to the nerve. Through this catheter, small quantities of local anesthetics can be continuously delivered for several hours after surgery, effectively relieving the worst of the pain.

To date, the administration of local anesthetics through a catheter next to the femoral nerve has been shown to improve pain relief after knee replacement surgery. These pain relief benefits have resulted in faster recovery after total knee replacement. Until recently, catheter techniques were not frequently used due to technical difficulties encountered when attempting to find the femoral nerve, as well as difficulties related to catheter displacement after surgery. Due to recent improvements in nerve and catheter localisation, catheter installation has become easier, more precise and more reliable. However, the distance at which the catheter must be advanced next to the femoral nerve in order to provide the best pain relief remains unknown. Insertion distance could influence the initial quality and distribution of the freezing, its duration, or both. Therefore, this study is designed to compare two catheter insertion distances, in order to help determine which is best for pain relief after knee surgery.

Patients will be randomly assigned to the following groups:

* Group 1: 3 cm insertion
* Group 2: 7 cm insertion

The anesthesiologist will insert a catheter close to the femoral nerve, at the junction of the thigh and torso immediately before beginning of anesthesia for surgery. The usual medication will be used to make installation more comfortable. The exact location where the catheter will be put into place will be identified using an ultrasound machine. This device will allow the anesthesiologist to identify the various anatomical structures. A specially designed needle will be inserted next to the femoral nerve, and its position will be confirmed with a neurostimulator. Once the adequacy of needle position is confirmed, the anesthesiologist will introduce 3 cm(Group 1) or 7 cm (Group 2)of the catheter through the needle, and then will withdraw the needle. The catheter will be fixed in place to avoid displacement.

Patients will receive standard regional or general anesthesia for this type of surgery.

After surgery, pain will be assessed using a verbal numeric pain scale. A Patient Controlled Analgesia pump will be provided to the patients. In addition, all patients will receive local anesthetics through their femoral catheter for at least 24 hours after surgery, which will partially freeze the knee.

Patients will be asked to fill out a pain intensity measurement form using a 0-10 pain scale at 3, 6 and 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older undergoing major knee surgery.

Exclusion Criteria:

* Coagulopathy
* Pregnancy
* Allergy to local anesthetics
* Patient unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sensory block assessment | 24 hours after surgery

SECONDARY OUTCOMES:
Quality of pain relief | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Williams, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Canada (2):
  - CSSS Chicoutimi, Chicoutimi, Quebec
  - Centre Hospitalier de l'Université de Montréal (Hôpital Notre-Dame), Montreal, Quebec